CLINICAL TRIAL: NCT05550298
Title: Multi-Center Molecular Diagnosis and Host Response of Respiratory Viral Infections in Pediatric Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: St. Jude Children's Research Hospital (Other); Seattle Children's Hospital (Other); The Children's Hospital at Montefiore (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: VIPER; 7R01AI159684-02 (NIH); NCI-2022-08554 (Other: National Institute of Health)
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic Cell Transplant; Solid Organ Transplant; Respiratory Viral Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hematopoietic Cell Transplantation (HCT): Early and accurate diagnosis of respiratory viral infections (RVIs) in children and adolescents who have undergone HCT is important for improving outcomes. The investigators are doing this study to understand more about how RVIs affect children who receive a transplant.
- Solid Organ Transplant (SOT): Early and accurate diagnosis of respiratory viral infections (RVIs) in children and adolescents who have undergone SOT is important for improving outcomes. The investigators are doing this study to understand more about how RVIs affect children who receive a transplant.

SUMMARY:
The participants are being asked to take part in this clinical trial, a type of research study, because the participants are scheduled to receive or have recently received a hematopoietic cell transplant (HCT) or a solid organ transplant (SOT).

Primary Objective

To determine if pre-transplant screening for respiratory viral load predicts RVI within 1- year post-transplant among survivors.

Secondary Objectives:

* To develop and validate a classifier based on pre-transplant immunological profile predictive of developing an acute respiratory viral infection (aRVI), with RSV/PIV3/HMPV/SARS-CoV-2 through one-year post-transplant among survivors.
* To develop and validate a classifier based on Day +100 post-transplant immunological profiles predictive of developing an acute respiratory viral infection (aRVI),with RSV/PIV3/HMPV/SARS-CoV-2 through one-year post-transplant among survivors .

DETAILED DESCRIPTION:
The investigators will collect a nasal swab and blood sample from the participant when the participant is enrolled on the study and if the participant develops a RVI in the first year after transplant. The investigators will collect a blood sample 100 days after the participant's transplant.

ELIGIBILITY:
Recipient Inclusion Criteria

* Less than 18 years at the time of anticipated transplant
* Participant meets one of the following criteria:

  1. scheduled to receive allogeneic hematopoietic cell transplant within 14 days of enrollment or
  2. Scheduled to or received solid organ transplant within 7 days before or after enrollment
* Participant is receiving care at the time of enrollment at one of the study participating institutions.
* Parent/guardian willing and able to provide informed consent, and if appropriate, child willing and able to provide informed assent.

Donor Inclusion Criteria

* Donor for HCT recipient enrolled on the VIPER study.
* Willing and able to provide informed consent.

Exclusion Criteria:

Recipient Exclusion Criteria

None

Donor Exclusion Criteria

* Is not an HCT donor for a participant enrolled on the VIPER study.
* Not available to provide pre-transplant research blood sample.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants developing a RVI within one-year post transplant. | Baseline through 1-year post-transplant
  Prevalence is estimated as the proportion of HCT or SOT participants with a positive PCR pre-transplant screen who develop any RVI within one year post transplant. A 95% confidence interval will be provided.

SECONDARY OUTCOMES:
Predicted risk of a post-transplant recipient developing an aRVI within one-year post-transplant | 1 year
  Risk will be predicted by the development of a pre-transplant immunology model utilizing measurements of pre-transplant quantitative immunology (recipient and donor) and RSV/PIV3/HMPV/SARS-CoV-2 RVI from pre-transplant to year one post-transplant
Predicted risk of a post-transplant recipient developing an aRVI from Day 100 to one year post transplant. | Day +100 through 1-year post-transplant
  Risk will be predicted by the development of a pre-transplant immunology model utilizing measurements of Day 100 quantitative immunology (recipient and donor) and RSV/PIV3/HMPV/SARS-CoV-2 RVI from Day 100 to year one post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Maron, MD, Principal Investigator — St. Jude Children's Research Hospital; William J. Steinbach, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (27):
- United States (27):
  - University of Alabama at Birmingham's (UAB), Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's National Medical, Washington D.C., District of Columbia
  - University if Miami, Miami, Florida
  - Emory and Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Chicago Medicine Comer Children's Hospital, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Le Bonheur, Memphis, Tennessee
  - Cook Children's, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Center Center, Houston, Texas
  - UTHealth Houston, Houston, Texas
  - Seattle Childrens, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols